CLINICAL TRIAL: NCT04965974
Title: Efficacy of Blue Wavelength in Managing Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Shumaila Masood, Principal investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUF/MPO/2101
Record Dates: First submitted 2021-06-10; First posted 2021-07-16 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: The digital blue light blocking filter will be randomly installed in digital devices of the 80 subjects and rest of 80 will be without filter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 blue light blocking filter group (Experimental): digital blue light blocking filter is installed laptops and mobile phones of 80 individual using digital devices more than 4 hours. asked them to use the filter continuously while using digital devices.
  Interventions: Device: Digital blue light blocking filter
- 2 non filter users (Experimental): Effect of time duration of digital screen on the dry eyes is checked.
  Interventions: Device: Digital blue light blocking filter

INTERVENTIONS:
Device: Digital blue light blocking filter — digital blue light blocking filter will be given to 80 dry eye subjects in mobile phones and laptops and 80 individuals will be without filters digital devices users
  Other Names: F.lux and blue light filter Night mode,Night shift

SUMMARY:
The study is conducted to evaluate the efficacy of digital blue light blocking filter in improvement of clinical indices of dry eye and ocular symptoms related to dry eye.

Introduction: Dry eye disease is a multifactorial disease of the ocular surface caused by loss of tear film homeostasis resulting damage to the ocular surface and neurosensory abnormalities.

DETAILED DESCRIPTION:
60 subjects aged 20-35 years with ocular surface disease index score greater than 13 will be taken from the University of Faisalabad. After taking consent, procedure starts from history then Schirmer test 1 will be performed to measure the tear deficient dry eye. Tear break up time will be done to assess the evaporative dry eye. Corneal surface staining will be used to measure corneal erosions. OSDI questionnaire will be used for the evaluation of ocular symptoms related to dry eye. The digital blue light blocking filter will be randomly installed in digital devices of the 80 subjects and rest of 80 will be without filter. After baseline data follow ups will be after 3 weeks and second after 8 weeks of filter use. Schirmer test 1, tear break up time corneal surface staining and OSDI will be performed on both groups (filter users and non-filter users) for the evaluation of dry eye. Data will be analyzed using SPSS version 21. Result of this study will give knowledge that use of digital blue light blocking filters are useful in the management of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Females with age 20-35years
* using digital devices androids and laptops
* Ametropia of up to 1.0 Diopter sphere(DS) and astigmatism of less than 0.5
* Emmetropes.

Exclusion Criteria:

* Subjects using topical drugs
* Smokers
* Subjects undergoing dry eye treatment
* History of contact lens wear within the past three months
* Corneal surface disease other than dry eye
* Corneal or eyelid infections
* Corneal surgeries
* Refractive error of more than 1 DS of SE and astigmatism of greater than0.5DC
* Age <18 and >3 years
* Subjects already using blue light blocking filters
* I phone users
* Pregnant women
* Males

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The tendency of dry eye disease is more in females .
Enrollment: 160 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
tear break up time | 8 weeks
  improvement in evaporative dry eye will be assessed by improvement in tear break up time in seconds after filter use.
Schirmer test values | 8 weeks
  improvement in aqueous deficient dry eye by Schirmer test values in mm .
corneal surface staining | 8 weeks
  'corneal surface staining grade scale' assess the improvement corneal surface erosions after filter use

SECONDARY OUTCOMES:
ocular surface disease index questionnaire | 8 weeks
  improvement in ocular surface disease index score.13-22ocular surface disease index score mild dry eye ,23-32 score means moderate dry eye and ocular surface disease index greater than 33 indicate severe dry eye .

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Faisalabad, Faisalābad, Punjab Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No